CLINICAL TRIAL: NCT04501263
Title: Developing an Testing an Educational Intervention for the Management of Constipation for People With Advanced Cancer: a Feasibility Intervention Study (DEMCON)
Brief Title: Educational Intervention for Management of Constipation
Acronym: DEMCON
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Queen's University, Belfast (Other); University of Bristol (Other); Marie Curie Hospice, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: 18NI0074; MCCC-RP-16-A20993 (Other Grant/Funding Number: Marie Curie UK)
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: DEMCoN Educational Intervention — Educational programme on constipation for Health care professionals in this clinical specialist palliative care

SUMMARY:
The overall aim of the study is to develop and test the feasibility and acceptability of a novel educational intervention for HCPs to help them manage constipation experienced by people in the hospice setting. This stage aims to establish the feasibility of, and to pilot, a novel educational intervention for HCPs. Additionally, it also originally aimed to test the feasibility of the chosen measures of change in patient care, however this was not undertaken. In order to achieve this aim, the objectives are to:

* Implement the educational intervention across Marie Curie sites.
* Evaluate the likely effectiveness of the educational intervention on the knowledge and self-efficacy of HCPs.
* Explore the feasibility and acceptability of the educational intervention with HCPs, and identify factors associated with feasibility/acceptability
* Explore the feasibility and acceptability of research procedures, and identify factors associated with feasibility/acceptability
* Examine the effect of contextual factors upon the implementation and sustainability of the educational intervention in the hospice.
* Examine the suitability of outcome measures for HCPs

DETAILED DESCRIPTION:
An incremental, multi-method approach was adopted, in line with the MRC Framework for complex interventions. Four prior data collection phases helped to inform the development of the educational intervention (a review of guidelines and a systematic review of the existing literature Muldrew et al 2018; a clinical case note review (McIlfatrick et al 2019) and qualitative findings from patients, caregivers and health professionals (Hasson et al 2019). The refinement of the intervention involved the project's fourth step (unpublished). This was the use of the Nominal Group Technique (NGT) with 39 HCPs to help identify priorities in the assessment and management of constipation. The findings from the NGT were further ratified by an international review group (n=19) on constipation management and care.

A mixed methods approach was undertaken to inform the development of the intervention and assess its impact. A small cohort, one-sample repeated measures design was used to assess the impact of the intervention on the knowledge of participants (health care professionals). Data collection was focused on three primary groups of HCPs; nurses, medics, and pharmacists. Qualitative data were collected after the intervention to assess the appropriateness of the intervention, the support in the specialist palliative care unit to complete it, the overall processes surrounding its implementation, and any impact that participants felt it had on practice. These data were gathered from focus groups (n=4) with 14 HCPs and nine telephone interviews with managers and senior staff in the SPC units. The intervention was delivered, and participants were recruited from five specialist palliative care inpatient units in the UK (Northern Ireland, Scotland, and England).

HCPS (nurses, medics, pharmacists) were invited to participate if they met the following inclusion criteria; (i) working in a clinical capacity in the SPC inpatient unit; (ii) involvement in the management of patients with constipation; (iii) over 18 years of age; and (iv) able to provide written consent in English. The educational intervention was advertised across sites through Research Leads, flyers and the identification of a "champion", in conjunction with senior staff. HCPs who met the inclusion criteria and were willing to participate could sign up via a webpage containing an information sheet, consent form, and information on how to access the education programme.

Intervention development and implementation processes Based on the findings from the previous stages, a 6-week, online, educational program was created with Syngery Learning an online learning management company, on constipation assessment and management. Each week of the program consisted of a short theoretical introduction to key aspects of constipation (assessment, prevention, non-pharmacological management, pharmacological management, opioid induced constipation, and bowel obstruction). This was supplemented with a quiz, link to practice activity, and a group discussion in an online closed group. Participant's study was largely self-directed and flexible. They could log in at any time during the 6-week data collection period to complete the activities. Managers of the specialist palliative care units were supportive of the educational program and assisted in the practical elements of running the course, including releasing staff from their workload to complete the required activities. Participants were encouraged to complete these activities during their work hours.

Data collection Measures were completed online at baseline and after completion of the educational intervention. Competency measures were the primary outcome of the study, linked to the NiCan Framework for Generalist and Specialist Palliative and End of Life Care Knowledge and Skills Framework. Participants completed a competency assessment tool extracted from the Competency and End of Life Care Competency Tool and the Knowledge and Self-Efficacy Survey. The intervention was implemented gradually, over two separate occasions, enabling learning from the first phase to be incorporated into the second phase.

Qualitative Data Collection Qualitative data were collected after the intervention to assess the appropriateness of the resource, the support within the SPC unit to complete it, the overall processes surrounding its implementation, and any impact that participants felt it had on practice. This used focus groups and telephone interviews with managers and senior staff within the specialist palliative care units . Participants taking part in were invited to participate if they met set inclusion criteria; (i) employed by hospice as HCP; (ii) previous experience working with patients receiving palliative care who suffer from constipation; (iii) over 18 years of age; and (iv) Willing to participant in the study and have provided informed consent.

Cost analysis Information was collected on the time spent by staff on the training resource, by staff type and by study centre. Staff time was valued using unit costs obtained from the Personal Social Services Research Unit Costs of Health & Social Care 2018.

ELIGIBILITY:
Inclusion Criteria:

* Working in a clinical capacity in the SPC inpatient unit
* Involvement in the management of patients with constipation.
* Over 18 years of age;
* Able to provide written consent in English.

Exclusion Criteria:

* Anyone who did not meet the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care professionals (nurses, medics, pharmacists)
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Study specific questionnaire | October 2018- January 2019
  To evaluate the feasibility of delivering an educational intervention in a specialist palliative care setting
Study specific questionnaire | October-2018-January 2019
  To evaluate the acceptability of delivering an educational intervention in a specialist palliative care setting

SECONDARY OUTCOMES:
Knowledge and self-efficacy survey | October 2018-January 2019
  To evaluate the impact of the intervention on the knowledge of participants
Focus group and telephone interviews | October 2018- January 2019
  To explore managers and staffs views on the appropriateness of the resource, the support to complete it and process surrounding implementation and any perceived impact on practice.
Personal Social Services Research Unit Costs of Health and Social Care | October 2018-January 2019
  To assess the resources used in the intervention on the knowledge of participants Assess the costs associated with providing the intervention
Competency and end of life care competency tool | October 2018-January 2019
  To evaluate the impact of the intervention on the knowledge (competency) of participants

CONTACTS AND LOCATIONS:
Overall Officials: Sonja McIlfatrick, PhD BA, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Newtownabbey, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: July 2020-July 2025

REFERENCES:
- [Background] Muldrew DHL, Hasson F, Carduff E, Clarke M, Coast J, Finucane A, Graham L, Larkin P, McCorry NK, Slater P, Watson M, Wright E, McIlfatrick S. Assessment and management of constipation for patients receiving palliative care in specialist palliative care settings: A systematic review of the literature. Palliat Med. 2018 May;32(5):930-938. doi: 10.1177/0269216317752515. Epub 2018 Feb 12. PMID 29431016
- [Background] McIlfatrick S, Muldrew DHL, Beck E, Carduff E, Clarke M, Finucane A, Graham-Wisener L, Larkin P, McCorry NK, Slater P, Hasson F. Examining constipation assessment and management of patients with advanced cancer receiving specialist palliative care: a multi-site retrospective case note review of clinical practice. BMC Palliat Care. 2019 Jul 15;18(1):57. doi: 10.1186/s12904-019-0436-3. PMID 31307441
- [Background] Hasson F, Muldrew D, Carduff E, Finucane A, Graham-Wisener L, Larkin P, Mccorry N, Slater P, McIlfatrick S. 'Take more laxatives was their answer to everything': A qualitative exploration of the patient, carer and healthcare professional experience of constipation in specialist palliative care. Palliat Med. 2020 Sep;34(8):1057-1066. doi: 10.1177/0269216319891584. Epub 2019 Dec 23. PMID 31868574